CLINICAL TRIAL: NCT07186569
Title: The Effect of Digital Interactive and Face-to-Face Peer Support on Medical Students' Clinical Skill Performance, Reflection Skills, and Retention of Clinical Skills
Brief Title: Effect of Digital Interactive and Face-to-Face Peer Support on Medical Students' Clinical Skill Performance, Reflection Skills, and Retention of Clinical Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Mustafa Onur Yurdal, Principal Investigator, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-YÖNP-0719
Record Dates: First submitted 2025-09-16; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Clinical Skills Education; Peer Support Interventions; Medical Students; Objective Structured Clinical Examination; Clinical Competence; Education, Medical, Undergraduate; Students, Medical; Social Support
Keywords: Peer support; Digital learning; Face-to-face learning; OSCE; Reflection; Skill retention; Medical students; Clinical skills; Randomized Controlled trial

STUDY DESIGN:
Intervention Model Description: Individually randomized, parallel-group, three-arm educational trial. Participants are allocated in a 1:1:1 ratio to: (A) Digital Interactive Peer Support, (B) Face-to-Face Peer Support, or (C) Standard Training (control). Interventions are delivered during the clinical skills course; there is no masking. Outcomes are assessed immediately post-intervention, with a follow-up assessment to evaluate retention at a predefined interval.
Who Masked: Outcomes Assessor
Masking Description: OSCE assessors were blinded to group assignment. Students were instructed not to disclose allocation, and assessment materials contained no arm-specific cues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Digital Interactive Peer Support (Experimental): Structured peer support via an online platform (modules, quizzes, discussion, and peer feedback).
  Interventions: Behavioral: Digital Interactive Peer Support
- Face-to-Face Peer Support (Experimental): Structured in-person peer sessions with guided practice, observation, and formative feedback (fece-to-face)
  Interventions: Behavioral: Face-to-Face Peer Support
- Standard Training (Usual Curriculum) (Active Comparator): Usual curriculum-based clinical skills training without additional structured peer support.
  Interventions: Behavioral: Standard Training (Control)

INTERVENTIONS:
Behavioral: Digital Interactive Peer Support — Individually randomized participants receive digital interactive peer support.
  Arms: Digital Interactive Peer Support
Behavioral: Face-to-Face Peer Support — Individually randomized participants receive face-to-face peer support.
  Arms: Face-to-Face Peer Support
Behavioral: Standard Training (Control) — Standard Training (Usual Curriculum)-Participants receive usual curriculum-based training without structured peer support.
  Arms: Standard Training (Usual Curriculum)

SUMMARY:
This randomized educational trial compares two peer-support approaches for teaching clinical skills to medical students. Participants are randomly assigned to one of three groups: (1) Digital interactive peer support delivered through an online platform with structured tasks and feedback; (2) Face-to-face peer support delivered in small group sessions with guided practice; or (3) Standard training according to the usual curriculum. All participants complete an objective structured clinical examination (OSCE) immediately after training, and complete a validated questionnaire to assess reflection skills. A follow-up OSCE is administered to evaluate retention of clinical skills. There is no drug or device involved and risks are minimal.

DETAILED DESCRIPTION:
Design: Interventional, randomized, parallel-assignment trial with three arms (digital interactive peer support, face-to-face peer support, standard training). Allocation is approximately equal across arms; masking is not used.

Setting and participants: Medical students who meet eligibility criteria at a university clinical skills program. Participants provide informed consent prior to enrollment.

Interventions:

* Digital interactive peer support - structured peer learning via an online platform (e.g., modules, quizzes, discussion, and peer feedback).
* Face-to-face peer support - structured in-person peer sessions with guided practice, observation, and formative feedback.
* Standard training - the usual curriculum without additional structured peer-support.

Assessments and timing: A baseline checklist may be collected as part of routine instruction. Primary endpoint is the OSCE total score obtained immediately post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled medical students [1st year]
* Age ≥18 years and able to provide informed consent
* Sufficient proficiency in the language of instruction
* Access to the digital platform (for the digital arm)
* Availability for post-intervention and follow-up assessments

Exclusion Criteria:

* Prior formal certification or extensive training in the targeted clinical skills
* Inability to attend scheduled peer-support sessions (digital or face-to-face)
* Conditions that would prevent participation in OSCE/assessment procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Objective Structured Clinical Examination (OSCE) Total Score | Immediately post-intervention
  Assessed using an OSCE comprising standardized stations scored with validated checklists. Total score range [min-max] points; higher scores indicate better clinical skill performance. No results or conclusions are included here.

SECONDARY OUTCOMES:
Reflection Skills Scale Total Score | Immediately post-intervention
  Assessed using a validated reflection skills instrument [write the full, unabbreviated scale name]. Scores range [min-max] points; higher scores indicate stronger reflection skills. No results or conclusions are included here.
Retention of Clinical Skills (OSCE Total Score) | 8 weeks post-intervention
  Follow-up OSCE total score at the specified time point using the same scoring rubric as the immediate OSCE. Higher scores indicate better performance. No results or conclusions are included here.

CONTACTS AND LOCATIONS:
Overall Officials: Remzi Yavas Kincal, PhD, Study Chair — Çanakkale Onsekiz Mart University
Locations (1):
- Faculty of Medicine, Çanakkale, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data. This study involves educational records and student assessment data; consent did not include external data sharing. Aggregate (de-identified) results will be available in publications.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT07186569/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT07186569/ICF_001.pdf